CLINICAL TRIAL: NCT02182388
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses (5 mg to 3000 mg) of BI 207127 NA as Powder in the Bottle Reconstituted With PEG 400/Tris/SDS in Healthy Male Subjects. A Randomised, Placebo-controlled and Within Dose Groups Double-blinded Trial. Followed by an Intra-individual, Partially Randomised, Open Comparison of Powder in the Bottle and Tablet Without and With Food.
Brief Title: Single Rising Oral Doses of BI 207127 NA as Powder in the Bottle in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241.1
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions

ARMS (3):
- BI 207127 NA (Experimental): single rising dose part
  Interventions: Drug: BI 207127 NA powder for solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 207127 NA, fasted or fed (Experimental)
  Interventions: Drug: BI 207127 NA powder for solution; Drug: BI 207127 NA tablet

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: BI 207127 NA powder for solution
  Arms: BI 207127 NA; BI 207127 NA, fasted or fed
Drug: BI 207127 NA tablet
  Arms: BI 207127 NA, fasted or fed

SUMMARY:
The objective of this trial was to investigate the safety, tolerability, pharmacokinetics, and relative bioavailability of BI 207127 NA as powder in the bottle (PIB) and solid oral dosage form (tablets) without and with food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥18 and Age ≤50 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nerve system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial.
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Inability to refrain from alcohol on trial days
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* Baseline prolongation of QTc interval >450 ms
* A history of additional risk factors for TdP (Torsades de points) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2007-01; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline, within 14 days after last trial procedure
Number of patients with clinically significant changes in vital signs (blood pressure (BP), pulse rate (PR) | Baseline, up to 14 days after last trial procedure
Number of patients with clinically relevant findings in 12-lead ECG (electrocardiogram) | Baseline, up to 14 days after last trial procedure
Number of patients with abnormal changes in clinical laboratory tests | Baseline, up to 14 days after last trial procedure
Number of patients with adverse events | up to 44 days
Assessment of tolerability on a 4-point scale by investigator | within 14 days after last trial procedure

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 72 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to the last observed plasma concentration) | up to 72 hours after drug administration
λz (terminal rate constant in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRToral (mean residence time of the analyte in the body after oral administration) | up to 72 hours after drug administration
CL/F (apparent clearance of the analyte in plasma after oral administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose) | up to 72 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 48 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 48 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 48 hours after drug administration